CLINICAL TRIAL: NCT00234416
Title: A Trial to Evaluate ZD1839 (IRESSA) in Combination With Radiotherapy & Gemcitabine as First-Line Treatment in Patients With Locally Advanced Pancreatic Cancer
Brief Title: IRESSA Combined With Radiotherapy & Gemcitabine as First-Line Treatment in Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0100
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; EGF-R
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gefitinib; Gemcitabine

INTERVENTIONS:
Drug: Gefitinib
Drug: Gemcitabine

SUMMARY:
The primary objective of the trial is to identify the dose of gemcitabine given as a 2-hour intravenous (iv) infusion that can be administered in combination with ZD1839 250 mg once daily and a standard course (45 Grays [Gy]) of radiotherapy in patients with locally advanced, unresectable pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed pancreatic cancer (aspiration biopsy by fine needle [PAAF] by USE or biopsy guide by ECO-CT). It is mandatory the diagnostic by USE and will recommend the aspiration biopsy with this technique
* Tumoural volume by TAC < 500 cc
* Aged 18 to 75 years inclusive
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) £ 1
* Life-expectancy of more than 12 weeks
* Women of child-bearing potential must be willing to practice reliable methods of birth control to prevent pregnancy

Exclusion Criteria:

* Previous radiotherapy or chemotherapy for malignant disease
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of basal cell carcinoma or cervical cancer in situ
* In the opinion of the investigator, any evidence of severe or uncontrolled systemic disease (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease)
* Absolute neutrophil count (ANC) less than 1.5 x 109/litre (L), platelets less than 100 x 109/L or haemoglobin less than 9 mg/dL; Prothrombin time (PT) less than 50%; Serum bilirubin greater than 2.5 times the upper limit of reference range (ULRR; Creatinine clearance less than 45 mL/min; ALT or AST greater than 2.5 times the ULRR
* Active dermatoses (e.g. psoriasis, eczema)
* Concomitant use of phenytoin, carbamazepine, barbiturates, rifampicin, or drugs with known corneal toxicity
* Known, severe hypersensitivity to ZD1839 or any of the excipients of this product

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2002-08; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Incidence of DLT

SECONDARY OUTCOMES:
Overall objective tumour response (CR and PR) based on the Response Evaluation Criteria in Solid Tumours (RECIST), assessed by abdominal CT (abdominal scan)
Nature, incidence and severity of adverse events (AEs) and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Spain Medical Director, MD, Study Director — AstraZeneca Spain
Locations (2):
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Valencia